CLINICAL TRIAL: NCT03310801
Title: Comparison of Clinical Outcomes Between Left Atrial Appendage Occlusion With Dual Antiplatelet Therapy Versus Conventional Antithrombotic Therapy in Patients With Atrial Fibrillation Undergoing Drug-eluting Stent Implantation
Brief Title: LAAO With DAPT Versus Antithrombotic Therapy
Status: Completed | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Severance Hospital (Other); Sejong General Hospital (Other); Gachon University Gil Medical Center (Other); Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cheol Woong Yu, Professor, Korea University Anam Hospital
Other Study IDs: LAAO with DAPT
Record Dates: First submitted 2017-09-17; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: left atrial appendage occlusion; antithrombotic therapy; atrial fibrillation; percutaneous coronary intervention; drug eluting stent
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LAAO with DAPT: patients with AF who underwent PCI and treated with LAAO(either ACP or Watchman) and DAPT
  Interventions: Procedure: ACP or Watchman
- Conventional antithrombotic therapy: patients with AF who underwent PCI and treated with conventional antithrombotic therapy

INTERVENTIONS:
Procedure: ACP or Watchman — Left atrial appnedage occlusion using ACP or Watchman
  Groups: LAAO with DAPT

SUMMARY:
This study will retrospectively review and compare clinical outcomes between left atrial appendage occlusion with dual antiplatelet therapy versus conventional antithrombotic therapy in patients with atrial fibrillation undergoing drug-eluting stent implantation.

DETAILED DESCRIPTION:
Composite of stroke and major bleeding will be compared after adjusting those groups using inverse probability weighted model.

ELIGIBILITY:
Inclusion Criteria:

* patients with AF who underwent PCI and treated with LAAO and DAPT or conventional antithrombotic therapy

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with AF who underwent PCI
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Composite of stroke and major bleeding | From date of index procedure until the date of primary endpoint occur or date of last follow up, whichever came first, assessed up to 50 months
  Primary endpoint is a composite of stroke and major bleeding. Stroke is defined as ischemic cerebrovascular event included both transient ischemic attack and ischemic cerebral infarction. Major bleeding event was defined as moderate or severe bleeding according to the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Woong Yu, MD, PhD, Principal Investigator — Korea University Anam Hospital

IPD SHARING:
Plan to Share IPD: Undecided